CLINICAL TRIAL: NCT06289595
Title: Impact of Photobiomodulation on Pain Associated With Orthodontic Treatment With Clear Aligners or Fixed Appliances - a Retrospective, Multicentered Study
Brief Title: Impact of Photobiomodulation on Pain Associated With Orthodontic Treatment
Status: Completed | Type: Observational
Sponsor: PBM Healing International Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00134382
Record Dates: First submitted 2024-02-22; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Orthodontic; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PBM: PBM = Use of PBM Ortho device
  Interventions: Device: PBM Ortho device
- Control: Did not receive any photobiomodulation treatment.

INTERVENTIONS:
Device: PBM Ortho device — Device emits light for photobiomodulation (light therapy).
  Groups: PBM

SUMMARY:
Orthodontic treatment can cause pain. Research studies have shown that light therapy can help reduce pain that is caused by orthodontic treatment. In this study, data was collected from the medical charts of patients who had orthodontic treatment and recorded their pain levels for 1 week at the beginning of orthodontic treatment while they used a light therapy device or did not use at device. This collected information was used to see if the light therapy device could lessen orthodontic pain.

DETAILED DESCRIPTION:
Orthodontic treatment can cause pain. This type of pain is the most common reason why patients stop orthodontic treatment or don't follow the instructions from the orthodontist. A company called PBM Healing has made a dental device called PBM Ortho that is used inside the mouth like a mouthguard. This device uses light therapy called photobiomodulation (PBM) to help with healing, move teeth faster, and lessen inflammation and pain. Other research studies have shown that light therapy can help reduce pain that is caused by orthodontic treatment.

In this research study, information from patients' medical charts was collected from 7 dental clinics located in Japan. Some patients at these clinics were asked to use the PBM Ortho device every day for 1 week and to record how much pain they were having. Other patients that did not use this device were simply asked to record their pain level every day for 1 week. This collected information was used to see if the light therapy device could lessen this pain from orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy male and female patients (age 18 - 65), i.e., did not suffer from systemic illness nor require medication during the study period.
* Permanent dentition, with Little's Irregularity Index (LII) of 2 mm or greater for the upper and lower arch.
* Orthodontic treatment using clear aligners or fixed appliances via non-extraction therapy.
* Non-smoker with no use of chewing tobacco.
* Good oral hygiene.
* Caries free.
* No sign of periodontal disease.

Exclusion Criteria:

* Systemic diseases
* Medication use for the past 6 months; especially use of anti-inflammatory (e.g., NSAIDs)
* Smoking.
* Active dental caries.
* Any periodontal problem including bleeding, tooth mobility, bone loss, attachment loss, deep pockets.
* Sleep apnea and other airway pathologies
* Photosensitivity or use of drugs that may cause photosensitivity
* Use of osteoporosis drugs
* Epilepsy
* Patients who had an implanted cardiac device unless the device is known to not be affected by magnetic fields

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that are 18-65 years old, both male and female, that are due to begin orthodontic treatment with either clear aligners or fixed appliances.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Level of Pain | 7 days
  Level of self-reported pain selected on a visual analog scale (VAS) form that rates pain level from 0 (no pain) to 10 (worst pain imaginable).

CONTACTS AND LOCATIONS:
Locations (7):
- Japan (7):
  - Bio Dental Clinic Ashiya, Ashiya
  - Sawa Dental Clinic, Kasugai
  - Soejima Dental Clinic, Kitakyushu
  - Higashimachigran Dental Clinic, Kumamoto
  - Tsujimura Dental Clinic, Tanabe
  - IXI Family Dental Clinic, Tokyo
  - Miki Dental Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: No